CLINICAL TRIAL: NCT02943837
Title: EUS-guided Fine Needle Aspiration (EUS-FNA) Versus EUS-guided Fine Needle Biopsy (EUS-FNB) for Diagnosis of Subepithelial Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kee Don Choi, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AMCSMT 001
Record Dates: First submitted 2016-10-20; First posted 2016-10-25 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Gastrointestinal Subepithelial Tumors

ARMS (2):
- EUS-FNA (Active Comparator): Device: 22G FNA needle
  Interventions: Procedure: Device: 22G FNA needle
- EUS-FNB (Experimental): Device: 20G FNB needle
  Interventions: Procedure: Device: 20G FNB needle

INTERVENTIONS:
Procedure: Device: 22G FNA needle
  Arms: EUS-FNA
Procedure: Device: 20G FNB needle
  Arms: EUS-FNB

SUMMARY:
Background: Preoperative pathologic diagnosis of subepithelial tumor (SET) can improve clinical decision making. Although EUS-guided fine needle aspiration (FNA) is currently considered the standard method for sampling SET, its diagnostic yield is generally suboptimal. EUS-guided fine needle biopsy (FNB) of SET is safe and feasible with adequate histology obtained.

Objective: To compare the diagnostic accuracy of EUS-FNA and EUS-FNB.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal, gastric, or duodenal SET over 2 cm
* Hypoechoic lesion including 4th layer on EUS

Exclusion Criteria:

* SET with characteristic findings such as lipoma, vessels, or ectopic pancreas
* bleeding or rupture of SET
* platelet count <50,000 or prothrombin time INR > 1.3

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy (proportion of correctly classified subjects (ture positive + true negative) among all subjects ) , compared to the gold standard diagnosis | 12 months
  Gold standard diagnosis is defined as;
  1. in operated patients; histological assessment of the surgical resection specimen
  2. in non-operated patients; based on the conclusions of the diagnostic work-up (combined outcomes of FNA and FNB samples and imaging studies)